CLINICAL TRIAL: NCT03192722
Title: Low Vision Patients' Preference for Colored Filters and Illumination for Near Reading Determined by the LuxIQ/2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Principal Investigator, So Yeon Lee, Assistant Professor, Nova Southeastern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-512
Record Dates: First submitted 2017-06-15; First posted 2017-06-20 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Ocular Conditions Resulting in Visual Impairment
Keywords: Filters; Illumination; Low vision; Reading
MeSH Terms: conditions — Vision, Low | interventions — Ultraviolet Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Immediate exposure to near vision glasses with filters (Experimental): Participants immediately provided with near vision glasses with colored filters
  Interventions: Device: Colored near reading glasses
- Delayed exposure to near vision glasses with filters (Other): Participants provided with near vision glasses with colored filters after 8 weeks of wearing clear near vision glasses
  Interventions: Device: Colored near reading glasses
- Immediate exposure to LuxIQ/2 (Other): Participants are examined with LuxIQ/2 to determine preferred lighting as determined by device followed by examination with OttLite Cobra
  Interventions: Device: Lighting as determined by LuxIQ/2 or OttLite Cobra
- Immediate exposure to OttLite Cobra (Other): Participants are examined with OttLite Cobra to determine preferred lighting followed by LuxIQ/2
  Interventions: Device: Lighting as determined by LuxIQ/2 or OttLite Cobra

INTERVENTIONS:
Device: Colored near reading glasses — Participants are provided with colored near vision glasses.
  Arms: Delayed exposure to near vision glasses with filters; Immediate exposure to near vision glasses with filters
Device: Lighting as determined by LuxIQ/2 or OttLite Cobra — Participants are provided preferred lighting (either OttLite or lamp with findings from LuxIQ/2)
  Arms: Immediate exposure to LuxIQ/2; Immediate exposure to OttLite Cobra

SUMMARY:
The effect of tinted filters and illumination on the visual performance of patients with low vision (i.e., individuals with reduced vision that is uncorrectable with glasses, surgery or treatments) has been a topic of research and discussion for many years, yet there is no current consensus or practice standard for the evaluation and recommendation of colored filters and/or illumination intensity. Anecdotally, there have been many subjective reports of improvement in visual function and comfort with the use of tinted lenses. Previous studies have attempted to elucidate the subjective improvements observed using vision tests, such as visual acuity and contrast sensitivity, and the findings have been inconsistent. Traditionally, filters and optimal illumination are prescribed clinically through a trial and error method, which involves trying various filters and lamps haphazardly to determine which if any are preferred by the patient. The investigators are proposing to evaluate whether the illumination and filters chosen in office by participants using a new assessment tool the LuxIQ/2 translate to overall patient comfort and improved speed, accuracy and print size while reading, and to evaluate whether participants have the same illumination and colored filter preference determined by the LuxIQ/2 in a clinical office setting and in their home environment. The investigators will evaluate whether participants prefer lighting determined by the new assessment tool the LuxIQ/2 in comparison to lighting determined by the OttLite Cobra in office.

DETAILED DESCRIPTION:
All eligible patients with complaints of difficulty performing sustained reading tasks, such as reading books or magazines, will be evaluated for their preference for filter color and lighting using the LuxIQ/2.

Baseline distance visual acuity, contrast sensitivity, and near visual acuity, will be evaluated during initial presentation to the clinic as part of usual care using validated tests that are routinely performed during a low vision examination. Best-corrected distance visual acuity will be determined using the ETDRS (Early Treatment for Diabetic Retinopathy Study) chart. Contrast sensitivity will be evaluated using the MARS contrast sensitivity chart. Best-corrected near visual acuity will be evaluated using the Lighthouse Continuous Text Card. The LuxIQ/2 will be administered 3 times at 15-minute intervals. Lighting preferences will be evaluated 3 times using the Ott Lite Cobra. Each subject will be asked to choose between their preferred lighting conditions as determined by the OttLite Cobra and the LuxIQ/2, i.e each participant ill choose which lighting conditions is preferred for reading. The assessment tool (OTTLite Cobra or LuxIQ/2) which is performed first will be randomized for each participant. Microperimetry (a type of visual field test) will be conducted on all participants using the MAIA microperimeter at the NSU site only.

For subjects who do not appreciate an improvement in reading ability with a colored filter in office, we will obtain their written informed consent to include data collected during the clinical examination. For participants who do not appreciate an improvement in reading ability with a colored filter, but who appreciate an improvement in reading ability with white light as determined by the LuxIQ/2 in comparison to the OttLite Cobra, appropriate light bulb and desk lanp will be provided as determined by the LuxIQ/2. For participants who prefer the lighting determined using the Ottlite Cobra, they will be provided with an Ottlite Cobra desk lamp as well as their preferred settings on the device as determined through the in-office evaluation to be used at home. Participants to whom light bulb recommendations were provided or the Ottlite Cobra was recommended to improve lighting for their reading tasks, will be contacted by a research assistant 1 week after the in office assessment to complete a telephone interview which will consist of an Activity inventory questionnaire which will inquire about their difficulty performing near tasks using their previous light source as well as Ramulu's sustained reading test. The Ramulu sustained reading test will be performed twice during the phone interview, once with their previous lighting they were using at home before they obtained the new reading lamp (where they do most of their reading) and again with their new desk lamp. After 1 month, the research assistant will call the participant to repeat the Activity questionnaire inquiring about ability to perform near tasks using the new recommended lighting.

For participants who appreciate an improvement in reading ability with colored reading glasses, we will obtain their written informed consent to join the longer-term study.

* Reading materials will be provided to participants in an enclosed envelope in office. Participants will be asked to refrain from opening envelope until contacted by research assistant. Other individuals who decide to participate at a later time after contemplating the requirements of the research, will be sent the reading material in the mail.
* A research assistant will contact subject 1 week after in office assessment to complete telephone interview which will consist of the reading domain of the Activity Inventory questionnaire and the modified Telephone Interview of Cognitive Status (TICS-M) and silent reading test. During the call, subject will be asked to read several pages of a short story to themselves, silently using their current reading glasses, not the new ones that will be ordered. Subjects will be asked to answer a few questions about the stories. This call should take about 30-60 minutes.
* Subjects will be provided with new prescription clear reading glasses. After 1 month a research assistant will contact participant to repeat the same questionnaires and silent reading test using a different short story.
* Within a month after the phone questionnaires, the PI will make an appointment to come to the subject's home to test near vision and contrast sensitivity and determine preference for filter in home environment. At this time, the PI may ask for the new pair of clear reading glasses to take them to our optical to tint the lenses to the color that is preferred by the subject.
* One group will obtain near vision glasses with color filter/tinted lenses immediately, while the other group (controls) will continue to wear the clear reading glasses for another 4 weeks and will then will crossover to obtain near vision glasses with the filter/tinted lenses.
* About a month after wearing near reading glasses with the colored lenses, one of our research assistants will call participant to repeat the same questionnaires and silent reading test again using a different short story. This call should take about 30-45 minutes.
* At the end a low vision optometrist on the research team will contact participants to ask some open-ended questions about what the participant thought about using the near reading glasses with the colored lenses. This call should take about 15-30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who express a desire to obtain filters in a pair of near reading glasses
* Age 18 and older
* Provide informed consent
* Complaints of difficulty performing sustained reading tasks, such as reading books or magazines
* Patients who are interested in obtaining preferred filters in a pair of reading glasses
* Patients who have completed an evaluation in the low vision service of the NSU The Eye Care Institute or Lighthouse of Broward or UCLA Stein Eye Institute

Exclusion Criteria:

* Subjects with a score less than 21 on the TICS-M
* Subjects diagnosed with Dry Eye Syndrome determined by clinical signs, history of or current topical prescription medication (i.e., Restasis or Xiidra) usage, or the usage of other dry eye treatment including punctal plugs, instillation of artificial tears more than once per day and advanced dry eye treatment
* Subjects with poor vision who would require electronic magnification or non-visual devices
* Patients with poor vision for whom clinical management strategy would not involve tinted reading glasses and a lamp

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Changes in Ramulu's sustained reading test | 12 weeks
  Measurement based on time taking to complete reading sections
Reading domain of Activity inventory | 12 weeks
  Measured based on scale of difficulty performing tasks

SECONDARY OUTCOMES:
Changes in near visual acuity | 12 weeks
  measured in M notation
Changes in contrast sensitivity | 12 weeks
  measured in log units

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Southeastern University, Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: No